CLINICAL TRIAL: NCT05516966
Title: A Phase 1, Randomized, Double-Blind, Placebo- and Positive-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous Injections of HRS9531 in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Subcutaneous Injections of HRS9531 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRS9531-102
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Intervention Model Description: HRS9531 injection compared with placebo and open positive-controlled group
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Participants receive low dose level of HRS9531 or matched placebo administrated by multiple subcutaneous injection
  Interventions: Drug: HRS9531; Drug: Placebo
- Group B (Experimental): Participants receive medium dose level of HRS9531 or matched placebo administrated by multiple subcutaneous injection
  Interventions: Drug: HRS9531; Drug: Placebo
- Group C (Experimental): Participants receive high dose level of HRS9531 or matched placebo administrated by multiple subcutaneous injection
  Interventions: Drug: HRS9531; Drug: Placebo
- Group D (Active Comparator): Participants receive Dulaglutide 1.5 mg by multiple subcutaneous injection
  Interventions: Drug: Dulaglutide Injection

INTERVENTIONS:
Drug: HRS9531 — Administrated SC
  Arms: Group A; Group B; Group C
Drug: Placebo — Administrated SC
  Arms: Group A; Group B; Group C
Drug: Dulaglutide Injection — Administrated SC
  Arms: Group D

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of multiple subcutaneous injections of HRS9531 in patients with type 2 diabetes mellitus who have suboptimal glycaemic control after conventional lifestyle or metformin intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Males and infertility females, 18-65 years of age, inclusive, on the date of signing informed consent.
2. Diagnosed with type 2 diabetes mellitus (T2DM) for at least 6 months.
3. Treated with conventional lifestyle intervention alone or stable treatment with metformin (≥1000 mg/day) at least 8 weeks prior to screening.
4. 7.0% ≤ HbA1c ≤10.5% at screening.

Exclusion Criteria:

1. History or presence of vital organ primary diseases, including but not limited to neuropsychiatric, cardiovascular, digestive, respiratory, urinary, endocrine, blood, immune and other diseases, judged by researchers to be unsuitable for this study.
2. Diagnosed or suspected with type 1 diabetes mellitus, special types of diabetes or secondary diabetes.
3. Have a history of acute complications of diabetes (diabetic ketoacidosis, lactic acidosis, hyperglycaemic hyperosmolar state, etc.) or episode of severe hypoglycaemic events within 12 months prior to screening.
4. Have a presence of proliferative diabetic retinopathy, diabetic macular edema, or nonproliferative diabetic retinopathy requiring treatment during the trial;
5. Participants in clinical trials of any drug or medical device in the 3 months prior to screening.
6. Breast-feeding women.
7. The investigator considers that the subject has any other factors that would make it inappropriate to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | Screening period up to Day 62
  A summary of adverse events, including serious adverse events (SAEs) and Hypoglycemic Events

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve (AUC) of HRS9531 | Start of Treatment up to Day 62
Maximum Concentration (Cmax) of HRS9531 | Start of Treatment up to Day 62
Change from Baseline in Fasting Blood Glucose (FBG) | Baseline up to Day 62
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline up to Day 29
Change from Baseline in Weight | Baseline up to Day 62
Immunogenicity: anti-HRS9531 antibody | Start of Treatment up to Day 62

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided